CLINICAL TRIAL: NCT02503865
Title: Phase 1-2 Study of Development of Rational Ways of Medical and Non-medical Treatment Methods for Metabolic Syndrome
Brief Title: Development of Rational Ways of Medical and Non-medical Treatment Methods for Metabolic Syndrome
Acronym: DRWMNTMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nazarbayev University (Other)
Collaborators: Institute Of Cardiology & Internal Diseases, Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Kuat Oshakbayev, Primary investigator, Nazarbayev University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0103RK00112
Record Dates: First submitted 2015-04-10; First posted 2015-07-21 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Diabetes mellitus,; Hypertension; Overweight; analimentary detoxication
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Hypertension; Overweight | interventions — Orlistat; Diltiazem; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional Patient group (Active Comparator): Xenical, Pionorm, Diroton, Diltiazem, Atorvastatin
  Interventions: Drug: Xenical, Pionorm, Diroton, Diltiazem, Atorvastatin
- "Analimentary detoxication" Weight loss (Experimental): Vegetables and salt diet
  Interventions: Dietary Supplement: "Analimentary detoxication"
- Healthy people (No Intervention): 64 healthy people

INTERVENTIONS:
Drug: Xenical, Pionorm, Diroton, Diltiazem, Atorvastatin — Xenical (Orlistat) - 120 mg/day in integration of Pionorm (Pioglitazone hydrochlorid) - 30 mg/day, Diroton (Lizinopril) - 20 mg/day, Diltiazem - 90 mg/day, Atorvastatin (Liprimar) - 40 mg/day
  Other Names: Conventional Patient group
  Arms: Conventional Patient group
Dietary Supplement: "Analimentary detoxication" — Vegetable and salt diet
  Other Names: Experimental Patient group
  Arms: "Analimentary detoxication" Weight loss

SUMMARY:
Metabolic syndrome: aetiology, pathogenesis, diagnosis, clinical management and prognosis

DETAILED DESCRIPTION:
Purpose: To create the complex scientifically proved concept of Metabolic syndrome (МS) development based on elaboration of the new methods of clinical diagnostics of МS components and highly effective МS clinical management in comparative studying of clinical, laboratory and cost effectiveness.

Participants and methods: This clinical study included 351 adults (184 female) in the Scientific research institute of cardiology and internal diseases (Almaty, the Republic of Kazakhstan). Statistical analysis was performed using Microsoft Excel-2008 in updating Lapach, Chubenko et al (2000) and SPSS for Windows v.17.0.

ELIGIBILITY:
Inclusion Criteria:

* written consent form
* age> 25 years
* skinfold thickness > 0,7 cm BP> 130/85 mm Hg or a patient on antihypertensive medications fasting blood glucose > 6.1 mmole/L, or 2-hour postprandial glucose level > 11.1 mmole/L / or a patient with type 2 diabetes blood cholesterol > 5.6 mmole/L possibility of treatment > 6 months follow-up > 1 year

Exclusion Criteria:

* complete immobilization of a patient (paresis /paralysis)
* patients with severe concomitant diseases of the kidneys and (or) of the liver
* early post-operative condition
* mental illness
* pregnancy
* persons who are in prison
* persons who are in military Armed Forces

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2003-01; Primary Completion 2008-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tabynbayev Nariman, Professor, Study Director — Nazarbayev University
Locations (1):
- Republican Scientific Center for Emergency Medicine, Astana, Astana, Kazakhstan

REFERENCES:
- [Background] Penn L, White M, Lindstrom J, den Boer AT, Blaak E, Eriksson JG, Feskens E, Ilanne-Parikka P, Keinanen-Kiukaanniemi SM, Walker M, Mathers JC, Uusitupa M, Tuomilehto J. Importance of weight loss maintenance and risk prediction in the prevention of type 2 diabetes: analysis of European Diabetes Prevention Study RCT. PLoS One. 2013;8(2):e57143. doi: 10.1371/journal.pone.0057143. Epub 2013 Feb 25. PMID 23451166
- [Background] Berk KA, Buijks H, Ozcan B, Van't Spijker A, Busschbach JJ, Sijbrands EJ. The Prevention Of WEight Regain in diabetes type 2 (POWER) study: the effectiveness of adding a combined psychological intervention to a very low calorie diet, design and pilot data of a randomized controlled trial. BMC Public Health. 2012 Nov 23;12:1026. doi: 10.1186/1471-2458-12-1026. PMID 23176668
- [Result] Browning JD, Baxter J, Satapati S, Burgess SC. The effect of short-term fasting on liver and skeletal muscle lipid, glucose, and energy metabolism in healthy women and men. J Lipid Res. 2012 Mar;53(3):577-586. doi: 10.1194/jlr.P020867. Epub 2011 Dec 3. PMID 22140269
- [Derived] Oshakbayev K, Dukenbayeva B, Togizbayeva G, Durmanova A, Gazaliyeva M, Sabir A, Issa A, Idrisov A. Weight loss technology for people with treated type 2 diabetes: a randomized controlled trial. Nutr Metab (Lond). 2017 Jan 31;14:11. doi: 10.1186/s12986-017-0163-9. eCollection 2017. PMID 28163748

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Patient Group: Xenical (Orlistat) 120 mg a day for 6 months with antidiabetes, antihypertensive therapy
  Xenical (Orlistat): Xenical (Orlistat) - 120 mg/day, Pionorm (Pioglitazone hydrochlorid) - 30 mg/day, Diroton (Lizinopril) - 20 mg/day, Diltiazem - 90 mg/day, Atorvastatin (Liprimar) - 40 mg/day
- "Analimentary Detoxication": Dietary Supplement - Vegetable and salt diet. Weight loss program "Analimentary detoxication"
  "Analimentary detoxication": Vegetable and salt diet
Period: Overall Study
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" | Healthy People
Started | 70 | 269 | 66
Completed | 65 | 222 | 64
Not Completed | 5 | 47 | 2
Not completed — Moved out of area | 1 | 8 | 0
Not completed — Refused treatment | 4 | 39 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" | Healthy People | Total
Number analyzed (Participants) | 65 | 222 | 64 | 351
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 46.5 (13.6) | 47.4 (12.8) | 47.7 (12.3) | 47.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 116 | 34 | 184
  Male | 31 | 106 | 30 | 167

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Level
Description: Fasting blood glucose (FBG) (mmole/L) and Two-hour postprandial glucose (THPG) (mmole/L) were measured.
Time Frame: up to 12 weeks
Measure: Mean (Standard Error); unit: mmole/L
Groups:
- "Analimentary Detoxication" Weight Loss: Dietary Supplement - Vegetable and salt diet. Weight loss program "Analimentary detoxication"
  "Analimentary detoxication": Vegetable and salt diet
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" Weight Loss | Healthy People
Number analyzed (Participants) | 65 | 222 | 64
mmole/L
  Fasting blood glucose level | 6.05 (0.46) | 6.43 (0.36) | 4.58 (0.18)
  Two-hour postprandial glucose | 14.5 (0.28) | 14.6 (0.28) | 5.3 (0.14)

2. Primary Outcome: Systolic/ Diastolic Blood Pressures (mm Hg)
Description: Systolic and Diastolic Blood Pressures (mm Hg) was measured by manual/automatic tonometery
Time Frame: up to 12 weeks
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" Weight Loss | Healthy People
Number analyzed (Participants) | 65 | 222 | 64
mm Hg
  Systolic Blood Pressures | 151.2 (1.1) | 152.1 (1.1) | 121.1 (0.7)
  Diastolic Blood Pressures | 94.1 (0.7) | 96.9 (0.8) | 79.9 (0.5)

3. Secondary Outcome: Lipid Profile
Description: Blood sample for lipid profile (Cholesterol in mmole/L, High-density Lipoproteids in mmole/L, Triglycerides in mmole/L) was measured
Time Frame: up to 12 weeks
Measure: Mean (Standard Error); unit: mmole/L
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" Weight Loss | Healthy People
Number analyzed (Participants) | 65 | 222 | 64
mmole/L
  Cholesterol | 5.22 (0.18) | 5.35 (0.17) | 4.9 (0.14)
  High-density Lipoproteids | 0.76 (0.007) | 0.75 (0.004) | 1.22 (0.007)
  Triglycerides | 2.1 (0.18) | 2.2 (0.12) | 1.4 (0.09)

4. Secondary Outcome: Immunoassay Hormones in Blood
Description: Immunoassay Insulin in the blood (in nU/L) was investigated
Time Frame: up to 12 weeks
Measure: Mean (Standard Error); unit: nU/L
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" | Healthy People
Number analyzed (Participants) | 65 | 222 | 64
nU/L | 22.9 (1.1) | 23.2 (1.0) | 6.5 (0.3)

5. Secondary Outcome: Immunoassay Cortisole in Blood
Description: Immunoassay Cortisole in the blood (nmole/L) was measured
Time Frame: up to 12 weeks
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" | Healthy People
Number analyzed (Participants) | 65 | 222 | 64
nmol/L | 743.8 (6.9) | 751.2 (6.7) | 445.3 (5.3)

ADVERSE EVENTS:
Arm/Group | Conventional Patient Group | "Analimentary Detoxication" | Healthy People
Serious Adverse Events (participants affected / at risk) | 29/65 | 26/222 | 0/64
Other Adverse Events (participants affected / at risk) | 49/65 | 62/222 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Patient Group (N=65) | "Analimentary Detoxication" (N=222) | Healthy People (N=64)
Indigestions (Gastrointestinal disorders) | 29 (78) | 26 (26) | 0 (0) — diarrhea, itching, gastritis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Patient Group (N=65) | "Analimentary Detoxication" (N=222) | Healthy People (N=64)
hypertermia (General disorders) | 40 (160) | 62 (124) | 0 (0)
hypertension (Cardiac disorders) | 42 (164) | 26 (52) | 0 (0)

LIMITATIONS AND CAVEATS:
We acknowledge the randomized clinical trial have not a large sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes